CLINICAL TRIAL: NCT03336645
Title: A Phase 3, Multicenter, Open-label Study to Determine the Efficacy, Safety, and Pharmacokinetics of Buccally Administered MHOS/SHP615 in Pediatric Patients With Status Epilepticus (Convulsive) in the Hospital or Emergency Room
Brief Title: Open-label Study of Midazolam Hydrochloride Oromucosal Solution (MHOS/SHP615) in Children With Status Epilepticus (Convulsive) in a Healthcare Setting in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP615-301
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-06

CONDITIONS: Nervous System Diseases
Keywords: Seizure; Midazolam hydrochloride; Convulsive
MeSH Terms: conditions — Nervous System Diseases; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHP615 (Experimental): Participants will receive a single age-specific dose (approximately 0.25 to 0.5 milligram per kilogram [mg/kg] as midazolam) of SHP615 oromucosal solution through buccal route upon onset of seizures.
  Interventions: Drug: SHP615

INTERVENTIONS:
Drug: SHP615 — SHP615 oromucosal solution will be administered as a single age-specific dose (2.5, 5, 7.5 and 10 mg).
  Other Names: Midazolam hydrochloride oromucosal solution; MHOS

SUMMARY:
The purpose of this study is to assess the efficacy, safety and pharmacokinetics of MHOS/SHP615 administered buccally in children with status epilepticus (convulsive) in a healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants whose corrected gestational age is greater than or equal to (>=) 52 weeks (gestational weeks plus the number of weeks after birth) and less than (<) 18 years (and weight greater than [>] 5 kilogram [kg]), at the time of investigational product administration. If the participant's exact age is not known, the participant should be excluded.
* Parent, guardian, or legally authorized representative (LAR) of the child provides informed consent (and assent, when applicable per Shire policy and country regulations) to participate in the study prior to participation in any protocol specific procedures. The participant may be prescreened by the investigator in their clinical practice and the parent, guardian, or LAR may sign informed consent before the participant presents to the healthcare setting for treatment of the seizure.
* Participant with generalized tonic-clonic SE with seizures accompanied by loss of consciousness with any of the following characteristics persistent at the time of study drug administration:

  1. Currently presenting with seizure (convulsive) activity and 3 or more convulsions within the preceding hour
  2. Currently presenting with seizure (convulsive) and 2 or more convulsions in succession without recovery of consciousness
  3. Currently presenting with a single seizure (convulsive) lasting >=5 mins

Exclusion Criteria:

* Female participants who are pregnant, suspected to be pregnant, or nursing.
* Subjects with major trauma, not necessarily restricted to the head, as the cause of the seizure.
* Subjects with seizures due to illegal drug or acute alcoholic intoxication.
* Subjects with known or suspected recurrent seizures due to illegal drug or alcohol withdrawal.
* Subjects with history of seizures of psychogenic origin.
* Subjects with seizures due to severe encephalitis or meningitis, as determined by the PI
* Subjects with known history of hypersensitivities, non-responsiveness or contraindications to benzodiazepines (ie, clinically significant respiratory depression, severe acute hepatic failure, myasthenia gravis, syndrome of sleep apnea, glaucoma with closed angle, use of concomitant drugs determined by the investigator to have a contraindication to the use of benzodiazepines.)
* Subjects with a known history of benzodiazepine abuse.
* Subjects who, in the judgment of the healthcare provider, have not responded to previous administrations of midazolam systemic therapies, including Midafresa and/or Dormicum.
* Subjects who need emergent surgical intervention and general anesthesia/intubation.
* Subjects with significant hypotension and cardiac dysrhythmia (example [eg], atrioventricular [AV] block of second or third degree, VT [ventricular tachycardia]).
* Subjects who have been receiving human immunodeficiency virus (HIV) protease inhibitors or HIV reverse transcriptase inhibitors.
* Subjects with current hypoglycemia (glucose <60 milligram per deciliter [mg/dL]) upon presentation at the hospital or healthcare setting.
* Subjects with severe cerebral anoxia (except cerebral palsy), in the judgment of the healthcare provider.
* Subjects have used an investigational product or been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
* Subjects has received antiseizure medication prior to arrival in the healthcare setting.
* Subjects has prior placement of a vagus nerve stimulator.

Ages: 3 Months to 216 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Study Physician, Study Director — Shire
Locations (23):
- Japan (23):
  - Yamanashi Prefectural Central Hospital, Kofu, Fujimi
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tokyo Women's Medical University Hospital, Tokyo, Kawadacho
  - NHO Minami-Okayama Medical Center, Okayama, Okayama-ken
  - Tokyo Women's Medical University Yachiyo Medical Center, Yachiyo, Owada Shinden
  - Jichi Children's Medical Center Tochigi, Saitama-shi, Saitama
  - Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Fukuoka Children's Hospital(NW), Fukuoka
  - NHO Hokkaido Medical Center, Hokkaidō
  - Kumamoto Saishunso National Hospital, Kumamoto
  - NHO Nagasaki Medical Center, Nagasaki
  - NHO Nishi Niigata Chuo National Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Nakano Children's Hospital, Osaka
  - Osaka Women's and Children's Hospital(NW), Osaka
  - Aichi Children's Health and Medical Center(NW), Ōbu
  - Saitama Children's Medical Center(NW), Saitama
  - Osaka University Hospital, Suita
  - National Center Hospital, NCNP, Tokyo
  - Tottori University Hospital, Tottori
  - Osaka University Hospital, Yamadaoka
  - Kanagawa Children's Medical Center(NW), Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Shire provides access to the de-identified individual participant data for eligible studies to aid qualified researchers in addressing legitimate scientific objectives. These IPDs will be provided following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.shiretrials.com website. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://www.shiretrials.com/en/our-commitment-to-transparency/data-sharing-with-researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 28 study centers in the Japan between 23 October 2017 (first participant first visit) and 19 August 2019 (last participant last visit).
Pre-assignment Details: A total of 25 participants were enrolled, received treatment and completed the study.
Groups:
- SHP615: Participants received single fixed age-specific dose (3 months to less than [<] 1 year received 2.4 milligram [mg]; 1 to < 5 years received 5 mg; 5 to <10 years received 7.5 mg and 10 to < 18 years received 10 mg) of midazolam hydrochloride oromucosal solution (MHOS) / SHP615 on Day 1.
Period: Overall Study
Arm/Group | SHP615
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who had received a single dose of the investigational product (IP), regardless of whether IP administration was documented to be complete or not on the IP administration page of the electronic case report form (eCRF).
Arm/Group | SHP615
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.63 (4.033)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response Rate
Description: Response rate was defined as the percentage of participants with therapeutic success. Therapeutic success was defined as the cessation of visible seizure activity within 10 minutes with a sustained absence of visible seizure activity for 30 minutes following a single dose of MHOS/SHP615 without the need for additional rescue medication.
Time Frame: From start of study drug administration up to 30 minutes post-dose
Population: Full Analysis Set (FAS) consisted of all participants in the safety set who had at least 1 assessment for determination of therapeutic success (date and time of the IP administration and seizure cessation for the initial seizure; participants with no recurrence of seizure within 30 minutes post-dose) performed after the administration of the IP.
Measure: Number; unit: Percentage of participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Percentage of participants | 80.0

2. Secondary Outcome: Percentage of Participants Who Had Sustained Absence of Seizure Activity for at Least 1, 4 and 6 Hours
Description: Percentage of participants whose seizure event stopped within 10 minutes of single dose administration of SHP615 and who had sustained absence of seizure activity for at least 1, 4, and 6 hours were reported.
Time Frame: From start of study drug administration up to 1, 4 and 6 hours post-dose
Population: FAS consisted of all participants in the safety set who had at least 1 assessment for determination of therapeutic success (date and time of the IP administration and seizure cessation for the initial seizure; participants with no recurrence of seizure within 30 minutes post-dose) performed after the administration of the IP.
Measure: Number; unit: Percentage of participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Percentage of participants
  Sustained Absence for at least 1 hour | 68.0
  Sustained Absence for at least 4 hours | 36.0
  Sustained Absence for at least 6 hours | 32.0

3. Secondary Outcome: Number of Participants With Time to Resolution of Seizures (Convulsions)
Description: Time to resolution of seizures (convulsions) was calculated as time from IP administration to the end of the initial seizure or administration of rescue anti-convulsant medication, whichever occurs first. Initial seizure referred to the seizure that triggered the use of the IP. Number of participants with time to resolution of seizures (convulsions) from the administration of SHP615 were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Participants | 21

4. Secondary Outcome: Number of Participants With Time to Recovery of Consciousness
Description: Time to recovery of consciousness (in minutes) was calculated only for participants who lost consciousness pre-dose at time from investigational product administration to recovery of consciousness post-dose or administration of rescue anticonvulsant medication, whichever occurs first. Number of participants with time to recovery of consciousness were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Participants | 19

5. Secondary Outcome: Percentage of Participants Who Required Additional Anticonvulsant Medication for Ongoing Status Epilepticus (SE)
Description: Percentage of participants who required additional anticonvulsant medication for ongoing SE, 10 minutes after a single dose of SHP615 were reported.
Time Frame: 10 minutes post-dose
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Percentage of Participants | 16.0

6. Secondary Outcome: Percentage of Participants Who Failed to Respond to the Treatment With SHP615
Description: Treatment failure/non-responder was defined as participants with continuing seizure activity and/or the need for any additional rescue medication according to the participating healthcare setting protocol or guideline, for 10 mins or more after a single dose of the IP.
Time Frame: 10 minutes post-dose
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Percentage of participants | 16.0

7. Secondary Outcome: Concentration of SHP615 in Plasma at 10 Minutes (C10)
Description: Concentration of SHP615 in plasma at 10 minutes were reported.
Time Frame: 10 minutes post-dose
Population: Pharmacokinetic (PK) set consisted of all participants who received a single dose of the IP and for whom at least 1 PK blood sample was collected post-dose. Here, the number of participants analyzed refer to the participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | SHP615
Number analyzed (Participants) | 16
nanogram per milliliter (ng/mL) | 45.2 (21.3)

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SHP615
Description: Cmax of SHP615 in plasma were reported.
Time Frame: 1, 3, 6 hours post-dose
Population: PK set consisted of all participants who received a single dose of the IP and for whom at least 1 PK blood sample was collected post-dose. Here, the number of participants analyzed refer to the participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SHP615
Number analyzed (Participants) | 16
ng/mL | 78.0 (16.4)

9. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 10 Minutes (AUC0-10) of SHP615 in Plasma
Description: AUC0-10 of SHP615 in plasma were reported. Here "min ng/mL" was minutes nanogram per milliliter.
Time Frame: Pre-dose, 10 minutes post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: min ng/mL
Arm/Group | SHP615
Number analyzed (Participants) | 16
min ng/mL | 304 (149)

10. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 60 Minutes (AUC0-60) of SHP615 in Plasma
Description: AUC0-60 of SHP615 in plasma were reported.
Time Frame: Pre-dose, 60 minutes post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: min ng/mL
Arm/Group | SHP615
Number analyzed (Participants) | 16
min ng/mL | 2965 (592)

11. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 180 Minutes (AUC0-180) of SHP615 in Plasma
Description: AUC0-180 of SHP615 in plasma were reported.
Time Frame: Pre-dose, 180 minutes post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: min ng/mL
Arm/Group | SHP615
Number analyzed (Participants) | 16
min ng/mL | 4411 (1140)

12. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of SHP615 in Plasma
Description: AUC(0-infinity) of SHP615 in plasma were reported.
Time Frame: Pre-dose, 1, 3, and 6 hours post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: min ng/mL
Arm/Group | SHP615
Number analyzed (Participants) | 16
min ng/mL | 5847 (2599)

13. Secondary Outcome: Time at Maximum Concentration (Tmax) of SHP615 in Plasma
Description: Tmax of SHP615 in plasma were reported.
Time Frame: 1, 3, and 6 hours post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: minutes
Arm/Group | SHP615
Number analyzed (Participants) | 16
minutes | 20.5 [15.5 to 28.0]

14. Secondary Outcome: Elimination Half-life (T1/2) of SHP615 in Plasma
Description: T1/2 of SHP615 in plasma were reported.
Time Frame: 1, 3, and 6 hours post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: minutes
Arm/Group | SHP615
Number analyzed (Participants) | 16
minutes | 115 [90.6 to 303]

15. Secondary Outcome: Number of Participants With Respiratory Depression
Description: Respiratory depression, included the following measures within 24 hours after administration of the IP: i) Persistent decrease in oxygen saturation to < 92 percent (%) measured at 10, 30 minutes, and 4, 6, and 24 hours post-dose (i.e, < 92 % on room air for 2 minutes or more after dosing while monitoring [per healthcare setting protocol and/or the clinical judgment of the physician]) ii) Increase in respiratory effort such that assisted ventilation is used (bag-valve-mask ventilation or endotracheal intubation). Number of participants with respiratory depression were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: Safety set consisted of all participants who had received a single dose of the IP, regardless of whether IP administration was documented to be complete or not on the IP administration page of the eCRF.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Participants
  Persistent Decrease in Oxygen Saturation | 0
  Increase in Respiratory Effort | 1

16. Secondary Outcome: Number of Participants With Aspiration Pneumonia Reported as Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs was defined as AEs that start or deteriorate on or after the date of the first dose of investigational product and no later than 3 days following the last dose of IP. Number of participants with aspiration pneumonia identified as TEAEs were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Participants | 0

17. Secondary Outcome: Change From Baseline in Riker Sedation-Agitation Scale at 24 Hours Post-dose
Description: Sedation-Agitation was assessed, using the "Riker Sedation-Agitation Scale" (SAS) by the following 7-point scale: 7. dangerous agitation; 6. very agitated; 5. agitated; 4. calm, cooperative; 3. sedated; 2. very sedated; 1. unarousable. Change from baseline in riker sedation-agition scale at 24 hours post-dose were reported.
Time Frame: Baseline, 24 hours post-dose
Population: Safety set consisted of all participants who had received a single dose of the IP, regardless of whether IP administration was documented to be complete or not on the IP administration page of the eCRF. Here, the number of participants analyzed refer to the participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | SHP615
Number analyzed (Participants) | 23
Score on the scale | 2.2 (1.23)

18. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs was defined as AEs that start or deteriorate on or after the date of the first dose of investigational product and no later than 3 days following the last dose of IP. Number of participants with TEAEs were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 25
Participants | 9

19. Secondary Outcome: Change From Baseline in Oxygen Saturation Percentage at 24 Hours Post-dose
Description: Oxygen saturation at baseline was measured and recorded on room air. The investigator had recorded the oxygen saturation, oxygen delivery system and amount of oxygen administered during the study. Change from baseline in oxygen saturation percentage at 24 hours post-dose were reported.
Time Frame: Baseline, 24 hours post-dose
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | SHP615
Number analyzed (Participants) | 14
Percentage of oxygen saturation | 3.7 (10.21)

ADVERSE EVENTS:
Time Frame: From start of study drug administration to follow-up (8 days).
Arm/Group | SHP615
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP615 (N=25)
Seizure cluster (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP615 (N=25)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (5):
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03336645/SAP_000.pdf
  • Study Protocol: Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03336645/Prot_001.pdf
  • Study Protocol: Amendment 1 (2017-07-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT03336645/Prot_002.pdf
  • Study Protocol: Amendment 2 (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT03336645/Prot_003.pdf
  • Study Protocol: Amendment 3 (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03336645/Prot_004.pdf